CLINICAL TRIAL: NCT06768281
Title: Comparison of the Efficacy of Lidocaine and Ozone in Masticatory Muscle Injections for Patients With Myofascial Pain
Brief Title: Effect of Lidocaine and Ozone in Injection for Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur Malkoc (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yağmur Malkoc, Assistant professor, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulMUH-DF-YM-02
Record Dates: First submitted 2024-12-19; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain Syndromes
Keywords: ozone; lidocaine; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streaming of patients and administration of substances (Experimental): 60 patients with myofascial pain syndrome who met the inclusion criteria were divided into four groups into isotonic saline, lidocaine, ozone gas and ozonated isotonic saline. Then the injections were done for each group.
  Interventions: Diagnostic Test: Headache Impact Test-6 (HIT-6); Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI); Diagnostic Test: Visual Analogue Score (VAS); Other: Masseter muscle injection
- Repetition of tests at certain intervals (Experimental): Quality of life was evaluated by administering PSQI and HIT-6 tests at postoperative 1st and 3rd months.
  Interventions: Diagnostic Test: Headache Impact Test-6 (HIT-6); Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI); Diagnostic Test: Visual Analogue Score (VAS)

INTERVENTIONS:
Diagnostic Test: Headache Impact Test-6 (HIT-6) — Patients who had injections were asked to mark their headache severities with a survey includes six questions about their past 4 weeks. The test applied preoperatively, postoperatively 1st and 3rd months.
Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI) — Patients who had injections were asked to reply some questions about their sleeping habits for past 4 weeks. The test applied preoperatively, postoperatively 1st and 3rd months.
Diagnostic Test: Visual Analogue Score (VAS) — Patients who had injections are asked to state their pain with a 10 cm visual analogue scale preoperatively and postoperatively 1st,2nd weeks and 1st and 3rd months.
Other: Masseter muscle injection — 1 ml of insulin needle with a 27-gauge ½ inch 13 mm needle tip will be injected into up to 4 trigger points in the taut bands that cause the most pain in the masseter muscle. Injections were done at most 3 times. As the control group, the first group was injected with isotonic saline; the second group was injected with 2% lidocaine without vasoconstrictor; the third group with ozone gas; and the fourth group with ozonated isotonic saline.
  Arms: Streaming of patients and administration of substances

SUMMARY:
Myofascial pain syndrome (MPS) is a chronic soft tissue rheumatism characterized by tense, painful muscle bands, known as trigger points, located within the muscle or fascia. These trigger points typically lead to pain during movement, limiting muscle extension and reducing mobility. While various treatments exist for MPS, the most common approach is injecting local anesthetic agents directly into the trigger points to relieve pain. Recently, systemic and local ozone therapy has also gained popularity as an alternative treatment for MPS. Ozone can be injected directly into muscles in areas such as the back and waist to target pain and inflammation. The aim of this study is to investigate the clinical effectiveness of ozone therapy with lidocaine injection in patients diagnosed with MPS.The aim of this study was to compare 2% non-vasoconstrictor lidocaine and ozone injections in the treatment of patients presenting to the clinic with myofascial pain syndrome and to determine the more therapeutic method.

DETAILED DESCRIPTION:
60 patients between the ages of 18-65 diagnosed with MPS were included in the study. The patients were randomly divided into four groups. As the control group, the first group was injected with isotonic saline, the second group was injected with 2% lidocaine without vasoconstrictor, the third group was injected with ozone gas and the fourth group was injected with ozonated isotonic saline. Patients were evaluated with VAS score before treatment, at 1, 2, 4 weeks and 3 months after treatment. In addition, quality of life was evaluated with HIT-6 and Pittsburgh Sleep Quality Index (PSQI) scales before treatment and at the 1st and 3rd months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* No temporomandibular joint treatment within the last year.
* Presence of palpable trigger points in the unilateral/bilateral masseter muscle.
* Classified as ASA 1 or ASA 2.
* Chronic pain in the masseter muscle for at least the past three months.
* Presence of at least two palpable trigger points in the unilateral or bilateral masseter muscle, with a pain score of ≥ 3 on the Visual Analog Scale (VAS) upon palpation

Exclusion Criteria:

* History of allergy to any anesthetic agent.
* Use of anticoagulant medications.
* Use of analgesics, muscle relaxants, or antidepressants within the last month.
* Diagnosed with specific conditions such as migraine, neuromuscular junction disorders, fibromyalgia, depression, or schizophrenia.
* History of trauma, tumor, or surgery in the head-neck region.
* Presence of skin infection in the relevant area.

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
1. The pain assessment after injections | Three months
  The primary outcome was the Visual Analog Score (VAS), a simple tool that allows the patient to express pain visually and numerically and is particularly effective in measuring subjective sensations. The patient is asked to choose a number between 0 and 10 indicating the pain level, with 0 indicating the least pain and 10 indicating the most pain.
2. Headache evaluation after injections | Three months
  The second outcome was the Headache Impact Test-6 (HIT-6), which is used to assess headaches. 6 indicates the lowest score, and 13 indicates the highest score.
3. Sleep quality evaluation after injections | Three months
  The third outcome was the Pittsburgh Sleep Quality Index (PSQI), consists of 7 main components and a total of 19 questions. Each component is scored from 0 to 3; the total PSQI score ranges from 0 to 21. High scores indicate a decrease in quality of life while descending scores indicate an increase.

CONTACTS AND LOCATIONS:
Overall Officials: ÇAĞRI DELİLBAŞI, PROF., Study Director — Medipol universitesi diş hastanesi
Locations (1):
- Istanbul Medipol University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albagieh H, Aloyouny A, Alshehri N, Alsammahi N, Almutrafi D, Hadlaq E. Efficacy of lidocaine versus mepivacaine in the management of myofascial pain. Saudi Pharm J. 2020 Oct;28(10):1238-1242. doi: 10.1016/j.jsps.2020.08.014. Epub 2020 Aug 28. PMID 33132718
- [Background] Yilmaz O, Sivrikaya EC, Taskesen F, Pirpir C, Ciftci S. Comparison of the Efficacy of Botulinum Toxin, Local Anesthesia, and Platelet-Rich Plasma Injections in Patients With Myofascial Trigger Points in the Masseter Muscle. J Oral Maxillofac Surg. 2021 Jan;79(1):88.e1-88.e9. doi: 10.1016/j.joms.2020.09.013. Epub 2020 Sep 14. PMID 33045182
- [Background] Kamanli A, Kaya A, Ardicoglu O, Ozgocmen S, Zengin FO, Bayik Y. Comparison of lidocaine injection, botulinum toxin injection, and dry needling to trigger points in myofascial pain syndrome. Rheumatol Int. 2005 Oct;25(8):604-11. doi: 10.1007/s00296-004-0485-6. Epub 2004 Sep 15. PMID 15372199
- See also: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/33132718/
- See also: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/33045182/
- See also: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/15372199/